CLINICAL TRIAL: NCT06598579
Title: Evaluation of the Effectiveness of Mindfulness-Based Cognitive Therapy for Depression, Implemented in Vietnamese Buddhist Pagoda
Brief Title: Evaluation of MBCT Implemented in Vietnamese Buddhist Pagoda
Acronym: MBCT-VN
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: VNU University of Education (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Bahr Weiss, Principal Investigator, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIHR21MH127563; R21MH127563 (NIH)
Record Dates: First submitted 2024-09-15; First posted 2024-09-19 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Depressive Symptoms; Quality of Life
Keywords: Depression; Mindfulness; Buddhist meditation; MBCT; Vietnam; task-shifting
MeSH Terms: conditions — Depression | interventions — Mindfulness-Based Cognitive Therapy

STUDY DESIGN:
Masking Description: Because a cluster-randomization design is being used, with random assignment at the pagoda-level to avoid cross-group contamination, masking is not possible.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MBCT-VN (Experimental)
  Interventions: Behavioral: Mindfulness-based Cognitive Therapy
- Buddhist Meditation - Treatment-as-Usual (Placebo Comparator)
  Interventions: Behavioral: Treatment-as-usual involving Buddhist meditation

INTERVENTIONS:
Behavioral: Mindfulness-based Cognitive Therapy — Mindfulness-Based Cognitive Therapy (MBCT) is a form of psychotherapy that combines principles of cognitive therapy with mindfulness practices focused on increasing non-judgemental awareness of the present moment. It was designed to help individuals, particularly those with depression, stop rumination and a cycle of negative thought patterns that lead to emotional distress including depression. It is a well established depression EBT. The Vietnamese version of the program (MBCT-VN) is a group treatment involving from five to ten participants (depending on how many participants are able to be recruited) per group.
  Other Names: MBCT
  Arms: MBCT-VN
Behavioral: Treatment-as-usual involving Buddhist meditation — MBCT and other mindfulness interventions were originally derived from Buddhist meditation, modifed to be non-secular and focused on treatment of depression and other mental health and behavioral problems rather than on spiritual development. In the present study, a treatment-as-usual condition involving Buddhist meditation will be used. The project will assess the characteristics of the Buddhist meditation delivered for the control group participants at pagoda meditation retreats but will not influence this control condition in any way.
  Arms: Buddhist Meditation - Treatment-as-Usual

SUMMARY:
Background

Depression presents a substantial public health burden around the world. Evidence-based psychotherapy treatments (psychotherapy EBT) for depression exist but access is often limited, particularly in low- and middle-income countries (LMIC), by mental health stigma and scarcity of professional mental health providers. One approach to address these issues is mental health task-shifting, transferring mental health services from highly trained mental health professionals operating in formal mental health settings, to non-mental health professionals or lay people receiving focused training in a particular mental health program, operating in non-mental health settings (e.g., schools; religious settings). Purposes of the present study are to (a) adapt Mindfulness-Based Cognitive Therapy (MBCT) for depression - a psychotherapy depression EBT - for implementation in Vietnamese Buddhist pagoda in VN (MBCT-VN); and (b) conduct a cluster-randomized clinical trial of MBCT-VN, implemented in Vietnamese Buddhist pagoda. Vietnamese Buddhist pagoda are selected as the task-shifting site because they represent a potentially low stigma, culturally-congruent site for task-shifting implementation of mindfulness-based mental health treatments.

Methods

MBCT was adapted for the present project through a collaborative team process, producing the MBCT-VN program. The clinical trial evaluation will involve a cluster-randomized comparison between (a) the treatment condition MBCT-VN, and (b) a treatment-as-usual control condition, Buddhist meditation as implemented in pagoda. To reduce cross-group contamination, pagoda will be the unit of assignment. Outcome assessments will include four timepoints across four months. One hundred and sixty adult participants will be recruited from eight (four treatment; four control) Buddhist pagoda in the Hanoi, Vietnam area. The primary outcome will be level of depression (Patient Health Questionnaire-9: PHQ-9); the secondary outcome will be quality of life (Quality of Life Enjoyment and Satisfaction Questionnaire: Q-LES-Q). The study will assess and evaluate several Implementation Science factors (e.g., Treatment Acceptability) as well as other potential moderators of treatment effects, and potential mediators such as increase in depression mental health literacy and decrease in depression stigma. Inferential analyses will use a general linear mixed model framework with a latent growth curve framework, with propensity covariates.

DETAILED DESCRIPTION:
Detailed Description

The study has three research aims and hypotheses:

* 1: To investigate the effects of MBCT-VN on the primary outcome, level of depression symptoms. It is hypothesized that the Treatment Group (MBCT-VN) will show significantly more reduction than the Control Group in PHQ-9 (depression) scores.
* 2: To investigate the effects of MBCT-VN on the secondary outcome, level of quality of life. It is hypothesized that the Treatment Group (MBCT-VN) will show significantly more increase than the Control Group in Q-LES-Q (quality of life) scores.
* 3: To investigate change from pre-treatment to post-treatment depression symptoms. It is hypothesized that the Treatment Group (MBCT-VN) will show pre-treatment to post-treatment change on the PHQ-9 that does not differ significantly from other within-group change in MBCT depression treatment evaluations, using statistical benchmarking methodology.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* PHQ-9 greater than or equal to 10
* PHQ-9 sadness item greater than or equal to 1, and / or PHQ-9 anhedonia item greater than or equal to 1

Exclusion Criteria:

* PHQ-9 greater than or equal to 20
* suicidal intent
* mania or psychosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2026-08-15 (Estimated); Study Completion 2026-10-15 (Estimated)

PRIMARY OUTCOMES:
PHQ-9 (Patient Health Questionnaire - 9) | From pre-treatment Baseline assessment (T1) , to 4 months post-baseline (T4) post-treatment follow-up
  This scale measures level of depression symptoms. Scores range from 0 to 27, with higher scores indicating higher levels of depression (worse outcome)

SECONDARY OUTCOMES:
Q-LES-Q (Quality of Life Enjoyment and Satisfaction Questionnaire) | From pre-treatment Baseline assessment (T1) , to 4 months post-baseline (T4) post-treatment follow-up
  This scale measures quality of life and functional impairment. Scores range from 13 to 65, with higher scores indicating higher levels of life functioning (better outcome).

CONTACTS AND LOCATIONS:
Locations (1):
- VNU University of Education, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Weiss B, Vu V, Dang HM, Trung L. Protocol for a cluster-randomized clinical trial to evaluate the effectiveness of mindfulness-based cognitive therapy for depression, implemented in Vietnamese Buddhist pagoda. BMC Psychol. 2025 May 20;13(1):527. doi: 10.1186/s40359-025-02754-5. PMID 40394634